CLINICAL TRIAL: NCT06960473
Title: A Prospective Randomized Controlled Clinical Study on Interventional Treatment of Budd-Chiari Syndrome Guided by IVUS and DSA
Brief Title: A Prospective Study on IVUS and DSA Guidance in the Treatment of Budd-Chiari Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XYFY2024-JS004-01
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Budd-Chiari Syndrome
MeSH Terms: conditions — Budd-Chiari Syndrome | interventions — Ultrasonography, Interventional; Angiography, Digital Subtraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVUS Group (Experimental): Patients receiving intervention guided by Intravascular Ultrasound (IVUS).
  Interventions: Device: Intravascular Ultrasound
- DSA Group (Active Comparator): Patients receiving intervention guided by Digital Subtraction Angiography (DSA).
  Interventions: Device: Digital Subtraction Angiography

INTERVENTIONS:
Device: Intravascular Ultrasound — In the IVUS group, the diameter of the reference vessel (the normal segment of the artery distal to the occlusion) is measured using Intravascular Ultrasound (IVUS). Based on the IVUS measurements, an appropriate balloon is selected to dilate the occluded segment.
  Arms: IVUS Group
Device: Digital Subtraction Angiography — The DSA group patients will have the appropriate balloon dilation selected for the occluded segment based on the DSA measurement results.
  Arms: DSA Group

SUMMARY:
This study aims to evaluate the effectiveness of interventional treatment guided by Intravascular Ultrasound (IVUS) compared to Digital Subtraction Angiography (DSA) in patients with Budd-Chiari Syndrome (BCS). Using a prospective, randomized controlled trial design, patients who meet the diagnostic criteria for BCS and are suitable for interventional treatment are randomly divided into the IVUS group and the DSA group. The IVUS group will undergo detailed assessment of vascular structure before interventional treatment to select the appropriate balloon for dilation, whereas the control group will make decisions based on DSA results. The primary endpoint of the study is the postoperative restenosis rate, while secondary endpoints include complications of interventional treatment, liver function, and patient survival rate. Successful implementation of this study will provide new technical means to optimize interventional treatment strategies for BCS, and help improve treatment outcomes and long-term prognosis for patients.

DETAILED DESCRIPTION:
This study aims to establish a precise interventional diagnostic and therapeutic system for Budd-Chiari Syndrome (BCS) based on IVUS assistance by comparing it with conventional DSA-guided diagnosis and intervention. The goal is to improve diagnostic accuracy and treatment outcomes for complex and difficult BCS patients using IVUS technology, reduce the incidence of postoperative restenosis, and enhance long-term patient prognosis. Specific objectives include:

1. Enhance the diagnostic accuracy for BCS patients, particularly in determining the nature of vascular obstruction and assessing hemodynamic status.
2. Optimize the interventional treatment strategy for BCS, including the selection and implantation of balloons and stents, and reduce surgical complications.
3. Increase the patency rate of vessels after interventional treatment and lower the incidence of restenosis.
4. Establish a set of IVUS-based precise diagnosis and treatment processes for BCS, promoting the application and dissemination of IVUS technology in BCS diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Primary Budd-Chiari Syndrome (narrowing or occlusion of the inferior vena cava near the hepatic veins or hepatic vein openings).
* Presence of membrane or short segment stenosis or occlusion suitable for balloon dilation (≤ 5 cm).
* Child-Pugh score less than 13.
* The patient or their authorized family member signs an informed consent form, voluntarily participating in the study and agreeing to follow-up.

Exclusion Criteria:

* Prior interventional treatment.
* Unfit for balloon dilation or stent placement (e.g., diffuse obstruction of the hepatic veins recommended for TIPS treatment, end-stage liver disease recommended for liver transplantation, etc.).
* Coexisting severe heart disease (such as heart failure, severe arrhythmias), liver or kidney failure, severe infections, iodinated contrast agent allergy.
* Coexisting hepatocellular carcinoma or other malignant tumors.
* Pregnant or breastfeeding women.
* Patients with a life expectancy of less than 1 year.
* Patients unable to complete follow-up or cooperate with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-05-18 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Restenosis | Follow-up and assessment will be conducted at 1 month, 3 months, 6 months, and 12 months post-surgery.
  At the 1 month, 3 months, 6 months, and 12 months follow-up after surgery, vascular patency will be assessed through imaging examinations such as ultrasound, CT, or MRI, and the incidence of restenosis will be recorded to compare the treatment outcomes between the IVUS group and the DSA group

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Interventional Radiology, the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China